CLINICAL TRIAL: NCT05205954
Title: HepHospital: A Pilot Trial of a Hepatology Home Hospital Intervention for Patients With Advanced Liver Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Nneka nnaoke Ufere, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021P002486
Record Dates: First submitted 2021-12-28; First posted 2022-01-25 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Cirrhosis; End Stage Liver DIsease; Liver Cirrhosis; Liver Disease Chronic
Keywords: Hospital at home; Home hospital
MeSH Terms: conditions — Fibrosis; End Stage Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hepatology Hospital at Home (Experimental): Patients with advanced liver disease receive hospital-level care in the home setting
  Interventions: Behavioral: Hepatology Home Hospital

INTERVENTIONS:
Behavioral: Hepatology Home Hospital — The Hepatology Home Hospital intervention entails the following: patient-reported symptoms and vital signs with appropriate triggers for phone calls and home visits, and regular communication with hepatology clinicians regarding care delivered at home to ensure continuity of care.

SUMMARY:
This research study is evaluating a program that entails a healthcare at home intervention for people with advanced liver disease.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥ 18 years old with diagnosis of cirrhosis based on histology, radiology, and/or elastography presenting to the emergency department or inpatient general medicine service
2. Patients must have one of the following:

   1. Ascites (requiring diuretics or serial large volume paracenteses)
   2. Hepatic hydrothorax (requiring diuretics)
   3. Hepatic encephalopathy (requiring medications)

Exclusion Criteria: All existing MGB home hospital criteria apply, with the following taking precedent for this specific condition

1. History of solid organ transplantation
2. On hemodialysis
3. MELD score > 20
4. Score <10 on Simplified Animal Naming Test (S-ANT1)
5. Current admission for hemodynamically significant GI bleeding or alcohol withdrawal
6. Require routine administration of controlled substances
7. Those deemed ineligible based on the MGH Home Hospital, inpatient medicine or hepatology clinician evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Escalation Rate | 18 months
  The intervention will be deemed feasible if less than 20% of enrolled patients have escalation of care back to the inpatient (brick-and-mortar) hospital

SECONDARY OUTCOMES:
Patient Experience | Up to 90 days
  To assess patient experience scores (Picker Patient Experience Questionnaire, Global satisfaction questionnaire) at discharge from HepHospital
Adverse Event Reporting | Up to 90 days
  We will assess rates of adverse events (acute kidney injury, falls, delirium, deep vein thrombosis/pulmonary embolism, escalation of care back to an inpatient hospital setting for at least 1 overnight stay, and death) for patient enrolled in HepHospital
Acceptability | 18 months
  Qualitative acceptability ratings from patients, caregivers, and clinicians obtained via exit individual interviews regarding acceptability (i.e. usefulness, effectiveness, and relevance of the intervention) from patients, family caregivers, and clinicians.

OTHER OUTCOMES:
Decline Rate | 18 months
  We will assess rates that patients decline to enroll in HepHospital
Quality of life (PROMIS-29 +2) | Baseline to post-discharge (+5 business day window) and 30-days (+10 business day window) post-discharge
  Change in participants' QOL as measured by the PROMIS-29+2 scale throughout the study.
Change in symptom Burden (Edmonton Symptom Assessment System-revised, ESAS-r) | Baseline to post-discharge (+5 business day window) and 30-days (+10 business day window) post-discharge
  Change in participants' symptom burden as measured by the ESAS-r throughout the study.
Unplanned readmission(s) after index hospitalization | Day of discharge to 30-days and 90-days post-discharge
  We will assess # of unplanned readmission(s) at 30- and 90-days post-discharge
Emergency Department Visit(s) after index hospitalization | Day of discharge to 30-days and 90-days post-discharge
  We will assess # of emergency department visit(s) at 30- and 90-days post-discharge
Total costs of care | 18 months
  To assess total costs of the acute care episode

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levine DM, Ouchi K, Blanchfield B, Saenz A, Burke K, Paz M, Diamond K, Pu CT, Schnipper JL. Hospital-Level Care at Home for Acutely Ill Adults: A Randomized Controlled Trial. Ann Intern Med. 2020 Jan 21;172(2):77-85. doi: 10.7326/M19-0600. Epub 2019 Dec 17. PMID 31842232
- [Background] Kahn-Boesel O, Mitchell H, Li L, Zhu E, El-Jawahri A, Levine D, Ufere NN. Hospital-Level Care at Home for Patients with Cirrhosis. Dig Dis Sci. 2024 May;69(5):1669-1673. doi: 10.1007/s10620-024-08361-5. Epub 2024 Mar 11. PMID 38466464